CLINICAL TRIAL: NCT06329479
Title: The RALI Study: a Multimodal Non-pharmacological (Clinical Review, Physical Activity, Bright Light Therapy and Cognitive Behavioural Therapy for Insomnia) Feasibility Trial for Circadian Rest-activity Rhythm Disorders in Patients With Advanced Cancer
Brief Title: A Feasibility Trial for Circadian Rest-activity Rhythm Disorders in Cancer (RALI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Prof Andrew Davies, Professor of Palliative Medicine, University of Dublin, Trinity College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1926B
Record Dates: First submitted 2023-11-02; First posted 2024-03-26 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Circadian Rhythm Disorders; Cancer
Keywords: circadian rest-activity rhythms; advanced cancer; feasibility trial; multi-modal
MeSH Terms: conditions — Chronobiology Disorders; Neoplasms | interventions — Cognitive Behavioral Therapy; Ultraviolet Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multi-modal intervention (Experimental): Single arm study receiving a multi-modal intervention
  Interventions: Behavioral: Cognitive behavioural therapy for Insomnia (CBT-I); Device: Bright Light Therapy; Behavioral: Individualised activity plan; Other: Clincial review

INTERVENTIONS:
Behavioral: Cognitive behavioural therapy for Insomnia (CBT-I) — A psychoeducational and evidence-based skills and strategies course for insomnia delivered online over four lessons through ThisWayUp. This will be completed during an 8-week feasibility trial.
Device: Bright Light Therapy — Daily bright light therapy for 30 minutes on waking delivered using the Lumie-L light box during an 8-week feasibility trial.
Behavioral: Individualised activity plan — An individualised activity plan is created at baseline and adjusted weekly aiming to increased daytime physical activity and reduce sedentary behaviours. The activity plan takes into consideration personal interests, perceived barriers to activity and develops an activity plan using Specific Measureable Achievable Realistic and Timely (SMART) goals. This will take place during an 8-week feasibility trial.
Other: Clincial review — Two clinical reviews will take place during an 8-week feasibility trial and consider uncontrolled symptoms, medication and blood test abnormalities which may impact on rest and physical activity levels

SUMMARY:
Circadian rest-activity rhythm disorders are common in patients with cancer, particularly in advanced disease. A recent international e-Delphi study has outlined recommendations for the assessment and reporting of the disorder and subsequently an observation study is underway assessing a cohort of patients with advanced cancer. Affected patients are eligible to enter a feasibility study assessing a non-pharmacological multi-modal intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Outpatient
3. Diagnosis of advanced cancer (locally advanced, incurable, metastatic)
4. Ambulatory
5. Estimated prognosis ≥ 3 months
6. Evidence of a circadian rest-activity rhythm disorder

Exclusion Criteria:

1. Inpatient
2. Engaged in shift-work
3. Long-haul travel in the last 14 days
4. Physical impairment limiting movement of the non-dominant arm
5. Cognitive impairment limiting the ability to complete the assessment tool and/or patient diary
6. Uncontrolled high blood pressure or tachycardia
7. Exercise-related symptoms and signs (e.g. chest pain, syncope, limb claudication, hypoxia at rest)
8. Participant has a history of uncontrolled mania or bipolar disorder
9. Participant has a recent history or current thoughts of self-harm or suicide
10. Participant has a recent change in antidepressant medication
11. Participant has an eye disorder (e.g. glaucoma, cataracts, retinopathy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
Acceptability and usability of a multi-modal non-pharmacological intervention | At the end of 8-weeks
  Patient completed questionnaire of the acceptability and usability of interventions and research assessments
Adherence to interventions | Outcome assessed weekly during the 8-week trial
  Patient completed weekly diary of adherence to the interventions and weekly monitoring by the researcher
Adverse events | Outcome assessed weekly during an 8-week trial
  Number of subjects develop adverse events during the trial in accordance with the Common Terminology Criteria for Adverse Events (CTCAE)
Completion rates of research assessments | Completed at baseline, week 2, week 4 and week 8
  Number of participants completing the midpoint and end of study assessments
Recruitment rate | 1 year
  Number of participants recruited to the feasibility study over a 1 year period

SECONDARY OUTCOMES:
Symptom assessment | Time 1 (baseline), Time 2 (end of 4 weeks), Time 3 (end of 8 weeks)
  Memorial Symptom Assessment Score Short Form (MSAS-SF). The scale assesses the presence and level of distress (Not at all, A little bit, Somewhat, Quite a bit, Very much) associated with 32 physical and psychological symptoms. Higher scores suggest increased symptomatology and increased distress
Quality of Life assessment | Time 1 (baseline), Time 2 (end of 4 weeks), Time 3 (end of 8 weeks)
  European Organisation for Research and Treatment of Cancer QLQ-C30. Participants rate 28 symptom and quality of life measures on a scale (1 = Not at all, 2 = A little, 3 = Quite a bit, 4 = Very much). Higher scores suggest a worser outcome. Participants also rate their overall health and quality of life on a scale 1-7 (1 = very poor, 7 = excellent).
Daytime Sleepiness | Time 1 (baseline), Time 2 (end of 4 weeks), Time 3 (end of 8 weeks)
  Epworth Sleepiness Scale. Participants rate the likelihood of falling asleep in 8 scenarios. Higher scores suggest increased daytime sleepiness
Sleep Quality | Time 1 (baseline), Time 2 (end of 4 weeks), Time 3 (end of 8 weeks)
  Brief Pittsburgh Sleep Quality Index (bPSQI). Participants complete 6 questions with higher scores suggesting poorer sleep quality.
Physical activity assessment | Continuous midweek 72-hour monitoring at baseline, Continuous midweek 72-hour monitoring during week 7
  Physical activity will be captured over a continuous 72-hour period using wrist and thigh accelerometry. Accelerometry devices collect activity counts during 1 minute periods (epochs).
Physical activity and sleep assessment | Continuous midweek 72-hour monitoring at baseline, Continuous midweek 72-hour monitoring during week 7
  A novel diary will be completed. Daytime physical activity will be assessed (level of tiredness, level of exertion, time spent during different activity intensities). Additional medication, smoking, caffeine and alcohol use will be documented. Nighttime sleep will also be assessed (time in bed, time to lights off, time to fall asleep, waking time, out of bed time, sleep quality).

CONTACTS AND LOCATIONS:
Locations (2):
- Ireland (2):
  - Our Lady's Hospice & Care Services, Dublin
  - St James's Hospital, Dublin